CLINICAL TRIAL: NCT06655194
Title: A Randomized, Open Label, Semi-replicate Crossover Pharmacokinetic Study to Compare the Bioavailability of a Single Oral Dose of Aspirin® 81mg Quick Chews® and a Single Oral Dose of Acetylsalicylic Acid 81mg Chewable Tablets for Testing of Bioequivalence Under Fasting Conditions in Healthy Adult Subjects
Brief Title: A Study to Learn if There is a Difference in the Blood Levels of Acetylsalicylic Acid When Taken as Different Chewable Tablets on an Empty Stomach by Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 22518
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Bioequivalence; Healthy Volunteers; Platelet Aggregation Inhibition
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator-test-comparator (Experimental): Participants will be randomly assigned to the treatment sequence "comparator-test-comparator" according to a computer-generated randomization list.
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE004465, UI1610477); Drug: Acetylsalicylic Acid (BAYE004465, UI1615160)
- Test-comparator-test (Experimental): Participants will be randomly assigned to the treatment sequence "test-comparator-test" according to a computer-generated randomization list.
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE004465, UI1610477); Drug: Acetylsalicylic Acid (BAYE004465, UI1615160)

INTERVENTIONS:
Drug: Acetylsalicylic Acid (Aspirin, BAYE004465, UI1610477) — Chewable tablet, 81mg, oral
Drug: Acetylsalicylic Acid (BAYE004465, UI1615160) — Chewable tablet, 81 mg, oral

SUMMARY:
In this study, researchers want to learn if 2 different forms of acetylsalicylic acid (ASA) chewable tablets will have the same effect in the body. For this, they compared the blood levels of a new form of ASA chewable tablet, which is manufactured at a different site, with an approved ASA chewable tablet, on an empty stomach in healthy participants. This is done as part of the regulatory requirement for the marketing approval of the new ASA chewable tablet.

The study treatment, ASA, is an antiplatelet drug. It works by making the blood thinner and stopping the blood from clotting.

In this study, participants will be healthy and will not benefit from taking ASA chewable tablets. However, the study will provide information on how the new ASA chewable tablet, which is manufactured at a different site, has an effect on the body.

The main purpose of this study is to compare blood levels of the new ASA chewable tablet with the approved ASA chewable tablet when taken as a single dose on an empty stomach.

For this, the researchers will analyze:

* Area under the curve (AUC): a measure of the total amount of ASA in participants' blood over time
* Maximum observed concentration (Cmax): the highest amount of ASA in participants' blood after a single dose without food

This study will have 3 treatment periods of 4 days each. In each period, participants will take either the new or approved ASA chewable tablet on an empty stomach according to the order assigned to them. The 2 treatment sequences in this study are:

New chewable tablet, approved chewable tablet, new chewable tablet

Approved chewable tablet, new chewable tablet, approved chewable tablet

Each participant will be in the study for around 7 weeks, which includes:

* a visit within 21 days of the first period to confirm if the participant can take part in the study
* hospital stay of around 2 days in each period, during which, participants will take their assigned treatment, and have blood tests to check for drug levels
* a gap of 1 week after taking the treatment in each period

During the study, the doctors and their study team will:

* measure the level of the study treatment by taking blood samples
* check participants' health by performing urine tests, checking vital signs and checking heart health using an electrocardiogram (ECG)
* ask the participants questions about how they are feeling and what adverse events they are having

An adverse event is any medical problem that a participant has during a study. The study doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatment.

As this study is conducted in healthy participants who will not benefit from the treatment, access to the treatment after the study is not planned.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Healthy, ambulatory male and female subjects between 18 to 55 years of age the health status will be assured by a complete physical examination, medical history, Electrocardiogram (ECG), vital sign measurement, and clinical laboratory testing.
* Subjects with a body weight of at least 50 kg and a Body Mass Index (BMI) between 18.0 to 27 kg/m2 according to Quetelet index.
* Subjects who have signed the authorization for clinical examinations (F-21 C) as well as the informed consent (F-07 C) before carrying out any procedure pertaining to the study.
* Subjects with legal capacity.
* Subjects understanding the nature, scope and risk/benefit of the trial and willing to adhere to the study procedures.
* Subjects presenting the following ranges of physiologic parameters at the selection visit: systolic blood pressure (seated) for 90 to 139 mm/Hg, diastolic blood pressure from 60 to 89 mg/Hg, heart rate between 50 and 100 beats per minute and respiratory rate between 14 and 20 breaths per minute.
* ECG, Hematic Biometry, Urinalysis, Biochemical Profile in normal reference ranges.
* The participants (women) agree to take the necessary measures to avoid conception during the entire study and up to two weeks after its end.
* Female subjects must present a negative result for pregnancy.
* Subjects have to present a negative result for the antibodies of hepatitis B and hepatitis C.
* Subjects have to present a negative result with respect to Anti-human immunodeficiency virus (HIV) 1 and Anti-HIV 2 antibodies.
* Subjects have to present a negative result with respect to venereal disease research lab (RPR) test.
* Subjects have to present a negative result with respect to drug abuse (amphetamines, cocaine, cannabis, benzodiazepines and barbiturates) performed during the selection process/beginning of each study period.
* Subjects have to present a negative saliva alcohol test result at the beginning of each study period.

Exclusion Criteria:

* Subjects with any finding of physical examination (including blood pressure, heart and respiratory rate, ECG, and body temperature [forehead]) outside of normal ranges and of clinical relevance.
* History of asthma, urticaria or allergic-type reactions after taking aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs).
* Severe heart failure.
* Subjects with a history of chronic or recurrent cardiovascular, renal, hepatic, muscle, metabolic, immunological, gastrointestinal (especially history of bleeding, chronic gastritis or peptic ulcers) including constipation, neurological problems (especially history of epileptic seizures), endocrine, hematopoietic or any type of anemia, asthma, mental illness or other organic abnormalities.
* Subjects with a muscle injury within a range of 21 days prior to the start of the study.
* Subjects with a hereditary problem of galactose intolerance, lactase deficiency, or glucose-galactose mal-absorption.
* Subjects who need any type of medication besides the study drug (exception: paracetamol up to 1 g/day).
* Subjects that have been exposed to drugs known as inductors or liver enzyme inhibitors or who have taken drugs which are capable of altering the urinary pH, like antacids with sodium bicarbonate, potassium citrate, diuretics, or any potentially toxic drugs within the 30 days prior to the beginning of the study.
* Subjects who have received any prescribed or over-the-counter (OTC) drug product, including vitamins and herbal remedies 30 days (or 7 half-lives) prior to the beginning of the study.
* Subjects who have been hospitalized for any disorder within seven months prior to the beginning of the study.
* Subjects who received investigational products within 90 days prior to the study.
* Subjects with a known hypersensitivity to any of the ingredients of the test or reference formulation.
* Subjects presenting a food allergy.
* Subjects who have consumed charcoal grilled nourishment 48 hours prior to the beginning of both study periods.
* Subjects consuming xanthine- and quinine-containing food and beverages and certain fruit juices such as grapefruit juice within 48 hours before investigational medicinal product (IMP) administration.
* Subjects having consumed alcohol within 48 hours before screening and within 12 hours before IMP administration (on Day -1 verified by saliva alcohol test).
* Smokers or currently consuming any type of tobacco product(s) including any smoking cessation nicotine-containing product within the previous three months (e.g., nicotine patch, nicotine gum).
* Subjects consuming xanthine excessively (more than 5 cups of coffee or equivalent beverages like energy drinks per day).
* Subjects who have donated or lost 450 mL or more blood within the 90 days prior to the beginning of the study.
* Subjects with a record of alcoholism and drug abuse, psycho-active substances or chronic medication during the previous 2 years.
* Subjects who require special diet for any reason, for example vegetarian diet.
* Subjects with any incapacity to understand the nature, purpose and possible consequences of the study.
* Subjects unwilling to follow study requirements and procedures.
* Subjects presenting a positive test for hepatitis B surface antigen test, anti hepatitis C, virus (Anti-HCV), or HIV-1/2 antibodies and HIV-1 p24-antigen.
* Subjects presenting a positive drug screen test or any history or suspicion of barbiturate, amphetamine, benzodiazepine, cocaine and cannabis.
* Subjects with any active disease, acute or chronic.
* Subjects with febrile or infectious illness within 1 week before screening.
* Subjects with any other disease or condition which could influence the metabolism of the drug (e.g., endocrine diseases).
* Subjects with any gastrointestinal complaints within 1 week before screening (gastrointestinal disorders including irritable bowel and gastrointestinal ulcer or bleeding).
* Subjects with a medical disorder, condition or history of such disorder or condition that could impair the subject's ability to participate or complete this trial in the opinion of the investigator.
* Subjects practicing sports excessively within 5 days before start of the treatment phase.
* Subjects with a complete body fungal infection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-04-06 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
AUC(0-tlast) of ASA | Baseline (pre-dose) and at 0.083, 0.166, 0.250, 0.333, 0.416, 0.500, 0.583, 0.666, 0.750, 0.833, 0.916, 1.00, 1.25, 1.50, 2.00, 3.00, 4.00, 4.50, 5.00, 7.00, 9.00, 12.00 and 24.00 hours post dose in each treatment period
  AUC(0-tlast): AUC from time 0 to the last data point > lower limit of quantitation (LLOQ)
Cmax of ASA | Baseline (pre-dose) and at 0.083, 0.166, 0.250, 0.333, 0.416, 0.500, 0.583, 0.666, 0.750, 0.833, 0.916, 1.00, 1.25, 1.50, 2.00, 3.00, 4.00, 4.50, 5.00, 7.00, 9.00, 12.00 and 24.00 hours post dose in each treatment period

SECONDARY OUTCOMES:
AUC of ASA and salicylic acid | Baseline (pre-dose) and at 0.083, 0.166, 0.250, 0.333, 0.416, 0.500, 0.583, 0.666, 0.750, 0.833, 0.916, 1.00, 1.25, 1.50, 2.00, 3.00, 4.00, 4.50, 5.00, 7.00, 9.00, 12.00 and 24.00 hours post dose in each treatment period
Ke of ASA and salicylic acid | Baseline (pre-dose) and at 0.083, 0.166, 0.250, 0.333, 0.416, 0.500, 0.583, 0.666, 0.750, 0.833, 0.916, 1.00, 1.25, 1.50, 2.00, 3.00, 4.00, 4.50, 5.00, 7.00, 9.00, 12.00 and 24.00 hours post dose in each treatment period
t1/2 of ASA and salicylic acid | Baseline (pre-dose) and at 0.083, 0.166, 0.250, 0.333, 0.416, 0.500, 0.583, 0.666, 0.750, 0.833, 0.916, 1.00, 1.25, 1.50, 2.00, 3.00, 4.00, 4.50, 5.00, 7.00, 9.00, 12.00 and 24.00 hours post dose in each treatment period
  t1/2: half-life associated with the terminal slope
tmax of ASA and salicylic acid | Baseline (pre-dose) and at 0.083, 0.166, 0.250, 0.333, 0.416, 0.500, 0.583, 0.666, 0.750, 0.833, 0.916, 1.00, 1.25, 1.50, 2.00, 3.00, 4.00, 4.50, 5.00, 7.00, 9.00, 12.00 and 24.00 hours post dose in each treatment period
  tmax: time to reach Cmax (in case of two identical Cmax values, the first tmax will be used)
Cmax of salicylic acid | Baseline (pre-dose) and at 0.083, 0.166, 0.250, 0.333, 0.416, 0.500, 0.583, 0.666, 0.750, 0.833, 0.916, 1.00, 1.25, 1.50, 2.00, 3.00, 4.00, 4.50, 5.00, 7.00, 9.00, 12.00 and 24.00 hours post dose in each treatment period
AUC(0-tlast) of salicylic acid | Baseline (pre-dose) and at 0.083, 0.166, 0.250, 0.333, 0.416, 0.500, 0.583, 0.666, 0.750, 0.833, 0.916, 1.00, 1.25, 1.50, 2.00, 3.00, 4.00, 4.50, 5.00, 7.00, 9.00, 12.00 and 24.00 hours post dose in each treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- IPharma, S.A. de C.V., Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/22518